CLINICAL TRIAL: NCT04868487
Title: Effectiveness of Health Literacy Education for Nursing Students in Turkey
Brief Title: Effectiveness of Health Literacy Education
Acronym: HL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşegül Akca (Other)
Responsible Party: Sponsor-Investigator, Ayşegül Akca, Research Assistant, Ankara Yildirim Beyazıt University
Organization: Ankara Yildirim Beyazıt University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2018-455
Record Dates: First submitted 2021-04-24; First posted 2021-05-03 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Health Literacy Level
Keywords: health literacy; nursing education; undergraduate student; education

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The intervention group received four weekly training sessions of health literacy education. Each educational session lasted an average of 50 minutes. The students were divided into four groups with an average of 25 students in each group.
  Interventions: Other: Health Literacy Education
- Control (No Intervention): The control group had no educational interaction with the researcher after the pre-test. The control group was administered the one-week and three-month posttest THLS-32 by the researcher simultaneously with the intervention group.

INTERVENTIONS:
Other: Health Literacy Education — Health literacy education, consisting of four sessions, was given to the intervention group.
  Arms: Intervention

SUMMARY:
To determine the effect of health literacy education given to nursing students. The study was conducted at two university nursing departments in Turkey between December 2018 and March 2019. A total of 206 nursing students, 103 in the intervention and 103 in the control group, were included in the study. Health literacy education, consisting of four sessions, was given to the intervention group.

ELIGIBILITY:
Inclusion Criteria:

* Inadequate (0-25 points) health literacy level
* Problematic-limited (25-33 points) health literacy level
* Accepting to participate in the research
* Accepting to participate in the research

Exclusion Criteria:

* Adequate (33-42 points) health literacy level
* Excellent (42-50 points) health literacy level
* Foreign language students with limited language proficiency
* Visual-hearing disability
* Having a neuropsychiatric disease

Ages: 18 Years to 32 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 206 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-05-15 (Actual)

PRIMARY OUTCOMES:
Health literacy level (the Turkey's Health Literacy Scale (THLS-32)) | before the implementation
  The level of health literacy was evaluated in four categories according to the score obtained: (0-25) points: inadequate health literacy, (> 25-33) points: problematic - limited health literacy, (> 33-42) points: adequate health literacy, and (> 42-50) points: excellent health literacy. The health literacy level of the students was determined and the intervention and control group was selected from among the students with insufficient and problematic-limited health literacy level.
Health literacy level (the Turkey's Health Literacy Scale (THLS-32)) | one week after the implementation
  The health literacy levels of the students who received and did not receive the intervention were compared. The level of health literacy was evaluated in four categories according to the score obtained: (0-25) points: inadequate health literacy, (> 25-33) points: problematic - limited health literacy, (> 33-42) points: adequate health literacy, and (> 42-50) points: excellent health literacy.
Health literacy level (the Turkey's Health Literacy Scale (THLS-32)) | three months after the implementation.
  The health literacy levels of the students who received and did not receive the intervention were compared. The level of health literacy was evaluated in four categories according to the score obtained: (0-25) points: inadequate health literacy, (> 25-33) points: problematic - limited health literacy, (> 33-42) points: adequate health literacy, and (> 42-50) points: excellent health literacy.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Yıldırım Beyazıt University, Ankara, Çubuk, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Akca A, Ayaz-Alkaya S. Effectiveness of health literacy education for nursing students: A randomized controlled trial. Int J Nurs Pract. 2021 Oct;27(5):e12981. doi: 10.1111/ijn.12981. Epub 2021 Jun 1. PMID 34060169